CLINICAL TRIAL: NCT07280806
Title: Biopsychosocial Model-based Care Versus Routine Physical Therapy in Chronic Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Muhammad Tariq, Dr. Muhammad Tariq Shafi, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UOL/IREB/25/12/00010
Record Dates: First submitted 2025-11-19; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: Biopsychosocial model based care; Routine Physical therapy; Chronic Low back pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Biopsychosocial group) (Experimental): Participants allocated to the Biopsychosocial Model-Based Care group will receive a structured, multimodal physical therapy program that integrates physical, psychological, and social components of rehabilitation. The protocol is designed to address not only musculoskeletal impairments but also cognitive, emotional, and behavioral factors that influence chronic low back pain (CLBP).
  Each session will last approximately 45 minutes, conducted three times per week for the four weeks under the supervision of a licensed physiotherapist trained in the BPS approach.
  Interventions: Other: Biopsychosocial model based care
- Group B ( Routine Physical Therapy) (Active Comparator): Participants in the Routine Physical Therapy group will receive a standardized physical therapy program designed to address the physical and functional components of chronic low back pain (CLBP). This approach represents standard clinical practice focused primarily on pain reduction, muscle flexibility, and core stabilization, without formal incorporation of psychological or social interventions.
  Each treatment session will last 45 minutes, administered three times per week for the 4 weeks by a qualified physiotherapist.
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: Biopsychosocial model based care — Participants receive a multimodal physical therapy program integrating physical, psychological, and social dimensions of care.
  Each session lasts 45 minutes, conducted three times per week for the four weeks.
  The intervention includes:
  Baseline modalities: Electrical hot pack (10 min) and TENS (10 min, 80-100 Hz, 100 µs) for pain relief.
  Manual therapy: Maitland central postero-anterior mobilizations (Grade I-II, 3 × 60 s).
  Neural mobilization: Sciatic nerve slider, 2 sets × 10 repetitions. Exercise therapy: Abdominal bracing, gluteal activation, graded functional activities, progressed by FITT principles.
  Psychological education: Cognitive Behavioral Therapy (CBT) and Pain Neuroscience Education (PNE) modules targeting fear-avoidance beliefs, catastrophizing, and maladaptive pain perceptions.
  Guided imagery and relaxation: Short sessions for body awareness and movement confidence.
  Social component: Group exercise sessions (3 to 4 participants) to encourage peer interaction.
  Arms: Group A (Biopsychosocial group)
Other: Routine Physical Therapy — Participants in the control group will receive standard physical therapy for chronic low back pain, focusing on pain relief, flexibility, and core/lower limb strengthening. Each session lasts 45 minutes, three times per week for four weeks. Baseline modalities include an electrical hot pack (10 min) and TENS (10 min; 80-100 Hz, 100 µs). Stretching targets the hamstrings, glutei, iliopsoas, and lumbar extensors (20-30 s × 3-5 reps). Strengthening and stabilization involve abdominal bracing, gluteal isometrics, bridging, and planks, progressed per FITT principles (10-15 reps, 40-60% effort). Brief patient education covers ergonomics, posture, activity modification, home exercises, and strategies for managing flare-ups. No psychological or social interventions are included.
  Arms: Group B ( Routine Physical Therapy)

SUMMARY:
Chronic low back pain (CLBP) is a multifactorial condition influenced by physical, psychological, and social factors. Conventional physical therapy primarily targets biomechanical impairments, often neglecting psychosocial contributors that perpetuate chronic pain and disability. This randomized comparative clinical trial aims to evaluate the effectiveness of Biopsychosocial (BPS) model-based care versus routine physical therapy on pain, disability, psychosocial outcomes, and inflammatory response among adults with CLBP.

A total of ___ participants with CLBP (≥12 weeks) will be randomly allocated into two groups:

Routine Physical Therapy Group - receiving baseline hot pack and TENS, stretching (hamstring, gluteal, iliopsoas, and lumbar extensors), and strengthening/stabilization exercises (planks, abdominal bracing, gluteal isometrics, and bridging).

BPS Model-Based Care Group - receiving the same baseline treatment plus Maitland mobilization (Grade I-II central PA), sciatic nerve slider, abdominal bracing, graded functional activity, cognitive behavioral therapy (CBT), pain neuroscience education (PNE), guided imagery, and group-based functional exercise therapy.

Primary outcome measures include Pain Self-Efficacy, Oswestry Disability Index (ODI), and C-Reactive Protein (CRP). A secondary variable, Perceived Social Support, will assess the social component of recovery.

This study hypothesizes that the BPS model-based care will produce superior improvements in pain self-efficacy, functional disability, and inflammatory markers compared to routine therapy, supporting the integration of biopsychosocial rehabilitation in chronic low back pain management.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a complex and persistent condition with multifactorial origins involving physical, psychological, and social dimensions. Traditional physiotherapy management typically emphasizes biomechanical correction through exercises and modalities; however, recent evidence underscores the significant contribution of psychosocial factors-such as maladaptive beliefs, fear-avoidance behaviors, and low self-efficacy-in the persistence of pain and disability. The biopsychosocial (BPS) model of care integrates these dimensions to promote holistic recovery and long-term functional improvement.

This randomized comparative clinical trial aims to determine the effectiveness of BPS model-based care versus routine physical therapy on pain self-efficacy, disability, inflammatory status, and perceived social support in individuals with CLBP. A total of ___ participants meeting the inclusion criteria (age 25-60 years, pain duration ≥12 weeks) will be recruited and randomly assigned into two equal groups.

The Routine Physical Therapy Group will receive:

Baseline care: Moist hot pack and Transcutaneous Electrical Nerve Stimulation (TENS)

Stretching of hamstrings, glutei, iliopsoas, and lumbar extensors

Strengthening/stabilization: abdominal bracing, planks, gluteal isometrics, and bridging exercises

The BPS Model-Based Care Group will receive:

The same baseline treatment as the control group

Maitland mobilization (Grade I-II central posteroanterior)

Sciatic nerve slider

Abdominal bracing and graded functional activities

Cognitive Behavioral Therapy (CBT) sessions focusing on fear-avoidance and coping skills

Pain Neuroscience Education (PNE)

Guided imagery and group exercise therapy to enhance engagement and motivation

Interventions will be administered three times per week for 6 weeks under physiotherapist supervision.

Outcome Measures:

Primary outcomes will include Pain Self-Efficacy (PSEQ), Oswestry Disability Index (ODI), and C-Reactive Protein (CRP) as a biochemical indicator of systemic inflammation. Perceived Social Support (Multidimensional Scale of Perceived Social Support) will be evaluated as a secondary variable reflecting the social dimension of recovery.

Assessments will be conducted at baseline and after 6 weeks of intervention. Data will be analyzed using appropriate statistical tests to compare within- and between-group changes.

This study will provide evidence on the role of integrated biopsychosocial rehabilitation in improving physical, psychological, and social outcomes in chronic low back pain, potentially guiding future physiotherapy practice toward a more holistic model of patient-centered care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with non-specific chronic low back pain (pain persisting for more than 12 weeks).
* Pain intensity score of ≥3 on the Visual Analog Scale (VAS).
* Able to read and understand the study instructions and questionnaires (e.g., SF-36, Oswestry Disability Index).
* Not undergoing any current structured physiotherapy or psychological treatment specifically for low back pain.

Exclusion Criteria:

* o History of specific spinal pathology (e.g., spinal fracture, tumor, infection, or inflammatory diseases like ankylosing spondylitis).

  * Presence of neurological deficits (e.g., radiculopathy, cauda equina syndrome).
  * Previous lumbar spine surgery.
  * Current diagnosis of major psychiatric illness (e.g., severe depression, psychosis) that may interfere with participation.
  * Pregnancy or within 6 months postpartum.
  * Ongoing treatment with systemic corticosteroids or other medications affecting musculoskeletal health.
  * Participation in another clinical trial within the past 3 months.
  * Any other medical condition deemed by the investigator to contraindicate participation in the study.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline (pre-intervention), 4 weeks (post-intervention), and 8 weeks (follow-up)
  Measured using the Short-Form McGill Pain Questionnaire-2 (Short-Form McGill Pain Questionnaire Version 2), which evaluates sensory and affective dimensions of pain in individuals with chronic low back pain. The scale uses 22 items rated from 0 to 10, where 0 indicates "no pain" and 10 indicates "worst possible pain." The final score is the mean of all items, with higher scores representing worse pain. The instrument demonstrates excellent internal consistency (Cronbach's α = 0.89-0.91)
Inflammatory Marker (CRP) | Baseline (pre-intervention), 4 weeks (post-intervention), and 8 weeks (follow-up)
  C-Reactive Protein (C-Reactive Protein, CRP) will be measured in serum to assess systemic inflammation associated with chronic low back pain. Levels will be recorded in milligrams per liter (mg/L). Typical values range from 0 to 10 mg/L in healthy individuals, with higher values indicating greater systemic inflammation. High-sensitivity CRP (hs-CRP) assays with intra-assay coefficient of variation <10% will be used to ensure accuracy
Mental Health and well being | Baseline (pre-intervention), 4 weeks (post-intervention), and 8 weeks (follow-up)
  Evaluated using the Pain Self-Efficacy Questionnaire (Pain Self-Efficacy Questionnaire, which measures an individual's confidence in performing daily activities despite pain. The scale contains 10 items scored from 0 ("not at all confident") to 6 ("completely confident"), resulting in a total score range of 0 to 60. Higher scores indicate greater pain self-efficacy. The instrument demonstrates excellent reliability in musculoskeletal populations (Cronbach's α = 0.92)
Perceived Social Support | Baseline (pre-intervention), 4 weeks (post-intervention), and 8 weeks (follow-up)
  Perceived social support will be measured using the Multidimensional Scale of Perceived Social Support. This is a 12-item scale with responses scored on a 7-point Likert format ranging from 1 to 7, where 1 = Very strongly disagree and 7 = Very strongly agree.
  The total MSPSS score ranges from 12 to 84, and subscale scores (Family, Friends, Significant Others) range from 4 to 28. Higher scores indicate better (greater) perceived social support. The scale has demonstrated strong internal consistency, with Cronbach's alpha values 0.88-0.93.
Disability | Baseline (pre-intervention), 4 weeks (post-intervention), and 8 weeks (follow-up)
  Disability will be assessed using the Oswestry Disability Index , a 10-item questionnaire that measures functional limitations and activity restrictions related to chronic low back pain. Each item is scored on a 6-point scale from 0 to 5, giving a total possible score range of 0 to 50.
  The total score is then converted to a percentage (0%-100%), where higher scores indicate worse disability. The ODI demonstrates high reliability, with Cronbach's alpha values reported between 0.86 and 0.94.
Exercise Adherence | Baseline (pre-intervention), 4 weeks (post-intervention), and 8 weeks (follow-up)
  Exercise adherence will be measured using the Exercise Adherence Rating Scale. The Exercise Adherence Rating Scale consists of 6 scored items, each rated on a 5-point Likert scale from 0 to 4. The total score ranges from 0 to 24, with higher scores indicating better adherence to prescribed exercises (greater frequency, duration, and effort). The scale demonstrates good internal consistency, with reported Cronbach's alpha values ranging from 0.81 to 0.86

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Faiza Sharif, PhD, Study Director — University of Lahore; Prof. Dr shoaib waqas, PhD, Study Chair — Lahore University of Biological and Applied Sciences
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
baseline participants
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start Date: The de-identified individual participant data (IPD) and supporting information will be available after publication of the primary trial results, expected approximately 12 months after trial completion.
  End Date: Access will remain available for 5 years from the start date to qualified researchers who submit a formal request and agree to the data use terms.
Access Criteria: De-identified individual participant data (IPD) and supporting information will be available to qualified researchers for academic, non-commercial purposes. Researchers must submit a written request outlining the research objectives and intended use of the data. Requests will be reviewed by the principal investigator (Dr. Muhammad Tariq Shafi) and the institutional ethics committee to ensure appropriate use and participant privacy.
  Data Available:
  The shared dataset will include de-identified information on:
  Demographics (age, sex)
  Pain intensity (SF-MPQ-2)
  Disability (ODI)
  Pain self-efficacy (PSEQ)
  Perceived social support (MSPSS)
  Exercise adherence (EARS)
  Serum C-Reactive Protein (CRP) levels
  Supporting documents will include the study protocol, statistical analysis plan, and data dictionary to facilitate accurate interpretation.
  Access Method:
  Approved researchers will receive the dataset and supporting materials via secure institutional file transfer or password-protected